CLINICAL TRIAL: NCT01640028
Title: Exploratory Study of Intra and Inter-subject Variability in Sebum Excretion Rate
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Inno-6026
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Oily Skin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze the relationship between sebum excretion rate and the following factors:

* Hormone levels (testosterone, dehydroepiandrosterone sulfate)
* Expression of 5-α-reductase type 1 (a protein in sebaceous glands that transforms a hormone (testosterone) into another one that strongly stimulates sebum production)
* Diet
* Sun and ultraviolet light exposure.
* Facial washing routine
* Sleep patterns (time when you start sleeping and total sleep time)

This study will analyze the relationship between sebum excretion rate and the various factors that may influence it in approximately 40 subjects. It will be conducted in one center located in Montreal. All devices are known and have already been used in the past.

DETAILED DESCRIPTION:
A total of 40 subjects with a sebum excretion rate of at least 4 will be included. Subjects will be seen at Day 0 and Day 7. Casual sebum measurements will be performed at least 2 hours after washing the face in the morning with a Sebumeter® following a 30-second application of a Sebumeter® Measurement Cartridge to the forehead. Sebum excretion rates will be measured with Sebutape® applied to the right and left forehead at each visit. Each Sebutape® will be scanned and the area covered by sebum, seen as gray-black dots on the scanned Sebutape®, will be measured by an image analysis software. Circulating levels of free testosterone and DHEAS will be measured at each visit. A skin biopsy behind an ear will be performed at Day 0 and Day 7 to measure gene expression of the 5-α-reductase type 1. On Day 0 and Day 7, subjects will be required to take a 24-hour recall questionnaire. On Day 0 and Day 7, subjects will be questioned about the time of sleep induction, their total sleep time for the night preceding the visit, facial washing routine and the number of hours of direct and indirect UV exposure in the past 24 hours. On Day 0 and Day 7, subject's forehead skin temperature will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a sebum excretion rate of at least 4 at Day 0 on both sides of the forehead as measured with Sebutape.
2. Subject is 18 years of age or older at time of consent and is in generally good health.
3. Female subject is willing to use effective contraceptive method for at least 30 days before Day 0 and until the end of the study. Effective contraceptive methods are:

   1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
   2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
   3. Intrauterine device (IUD);
   4. Sterilization such as tubal ligation, oophorectomy, hysterectomy or vasectomized partner;
   5. Postmenopausal state for at least 1 year for female subject or female partner of male subject;
   6. Same-sex partner;
   7. Abstinence.
4. Subject has a negative urine pregnancy test at Day 0 visit for female subject of childbearing potential only.
5. Subject is capable of giving informed consent and the consent must be obtained prior to any study related procedures.

Exclusion Criteria:

1. Subject is currently pregnant or lactating.
2. Subject has any skin condition on the forehead that could interfere with sebum excretion measurement except for mild acne vulgaris.
3. Subject has received investigational drugs within the 28 days or 5 half-lives, whichever is longer, prior to Day 0 or plans to during the study period.
4. Subject has used any topical medication on the face within 14 days of Day 0 or plans to during the study.
5. Subject has applied cosmetics or emollients on the forehead the morning of Day 0 visit or plans to the morning of Day 7 visit.
6. At the investigator's discretion subject has current or history of alcohol or drug abuse that would interfere with the ability of the subject to comply with the study protocol.
7. Subject has used isotretinoin in the 52 weeks preceding Day 0 or plans to during the study.
8. Subject should not have swum in chlorinated water within 24 hours of the Day 0 visit or plans to within 24 hours of the Day 7 visit.
9. Known hypersensitivity/allergy to lidocaine
10. The subject has a history of keloids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 40 subjects, male or female, aged 18 years or older with a sebum excretion rate (SER) of at least 4 at Day 0 on both sides of the forehead as measured with Sebutape, will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intra subject variability of sebum excretion rate | 7 Days
  To study the relationship between intra-subject variability in sebum excretion rate and androgen levels, expression of 5-α-reductase type 1, diet, UV exposure and sleep patterns

SECONDARY OUTCOMES:
Inter subject variability in sebum excretion rate | 7 Days
  To study the relationship between inter-subject variability in sebum excretion rate and androgen levels, expression of 5-α-reductase type 1, diet, UV exposure and sleep patterns

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research
Locations (1):
- Innovaderm Research, Montreal, Quebec, Canada